CLINICAL TRIAL: NCT05091515
Title: Study of Thermoregulatory Reactions of the Body of Medical Workers Who Use Personal Protective Equipment From Biological Hazards
Brief Title: Thermoregulatory Reactions of Medical Workers Who Use Personal Protective Equipment From Biological Hazards
Status: Completed | Type: Observational
Sponsor: Federal State Budgetary Scientific Institution "Izmerov Research Institute of Occupational Health" (Other)
Responsible Party: Principal Investigator, Andrey Mikhailovich Geregey, Head of the Laboratory of Personal Protective Equipment and Industrial Exoskeletons, Federal State Budgetary Scientific Institution "Izmerov Research Institute of Occupational Health"
Other Study IDs: PPE-05
Record Dates: First submitted 2021-08-24; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Overheating
Keywords: Thermophysiology; Personal protective equipment from biological hazards; Medical workers; COVID-19; Working conditions
MeSH Terms: conditions — Sunstroke; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health workers: Medical personnel: doctors, nurses.
  Interventions: Other: Personal protective equipment from biological hazard

INTERVENTIONS:
Other: Personal protective equipment from biological hazard — Includes: isolation clothing, mask, eyewear, overshoes

SUMMARY:
This research will provide data on thermal condition, functional status and working conditions of medical workers who use personal protective equipment from biological hazards. Acquired data will be used to define acceptable period of use for these protective costumes.

DETAILED DESCRIPTION:
This research will recruit 14-20 volunteers. During 8 hours each subject will perform their work using protective costume. Heart rate, electrocardiogram, oxygenation, skin and air temperature under costume and hygrometric data will be registered. Also there will be questionnaires for volunteers for subjective assessment of thermal and moisture sensations and assessment of working conditions.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals (based on medical screening)

Exclusion Criteria:

* endocrinological diseases and disorders
* health deviations at the time of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Health workers
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Skin thermometry | 8 hours
  DS1923-F5 Thermochron iButtons ("MaximIntegratedProducts, Inc", USA)
Hygrometry under costume | 8 hours
  DS1923-F5 Thermochron iButtons ("MaximIntegratedProducts, Inc", USA)
Electrocardiography | 8 hours
  Electrocardiographic system "Poly-Specter-SM" (LLC "Neurosoft", Russia), all parameters.
Blood pressure | 8 hours
  Electrocardiographic system "Poly-Specter-SM" (LLC "Neurosoft", Russia)
Heart rate | 8 hours
  Electrocardiographic system "Poly-Specter-SM" (LLC "Neurosoft", Russia)
Breathing rate | 8 hours
  Electrocardiographic system "Poly-Specter-SM" (LLC "Neurosoft", Russia)
Air thermometry and hygrometry | 8 hours
  "METEOSCOP-M" (LLC "NTM-Zashchita", Russia)

SECONDARY OUTCOMES:
Oxygenation | 8 hours
  Pulse oximeter MD300C2 ("Choicemmed", China)

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Konyukhov, Principal Investigator — Junior scientist
Locations (1):
- Federal State Budgetary Scientific Institution Izmerov Research Institute of Occupational Health, Moscow, Russia